CLINICAL TRIAL: NCT03852550
Title: CHILD-BRIGHT READYorNot[TM] Brain-Based Disabilities Trial
Brief Title: READYorNot[TM] Brain-Based Disabilities Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The planned sample size was 264; 43 participants completed follow-up. With significant start-up delays and recruitment curtailed by the COVID-19 pandemic, the limited feasibility to recruit our sample ultimately led to the early stop of the trial.
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); The Montreal Children's Hospital Foundation (Unknown); McMaster Children's Hospital Foundation (Unknown); Hamilton Health Sciences Corporation (Other); New Brunswick Health Research Foundation (Other); The Hospital for Sick Children (Other); Harvard Medical School (HMS and HSDM) (Other); Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1666
Record Dates: First submitted 2019-02-19; First posted 2019-02-25 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2024-11

CONDITIONS: Autism Spectrum Disorder; Cerebral Palsy; Epilepsy; Fetal Alcohol Spectrum Disorders; Spina Bifida
Keywords: Health Care Transition; Brain-Based Disabilities; CHILD-BRIGHT; e-health application; randomized controlled trial
MeSH Terms: conditions — Autism Spectrum Disorder; Cerebral Palsy; Epilepsy; Fetal Alcohol Spectrum Disorders; Spinal Dysraphism

STUDY DESIGN:
Intervention Model Description: Embedded experimental model design, embedding a qualitative component within the randomized controlled trial (RCT). Randomization will be stratified by region with a 1:1 allocation ratio for patients: intervention group (receiving MyREADY Transition[TM] BBD App intervention) or control group (continuing with usual care). The unit of randomization is the patient, using variable block randomization with block sizes of 2, 4, 6 and 8.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care + MyREADYTransition[TM] BBD App (Experimental): Participants in the experimental Intervention group continue to get the same care they have been getting (their usual care) and they receive the MyREADY Transition[TM] BBD App e-health application. There are 19 parts in the App with videos and games to help youth learn and practice ways to manage their health. There are approximately 5-7 hours of content in total. Participants will be asked to wait at least one day between the parts. There is a timer in the App to help to moderate pace and align with how young people learn and digest information. Participants can choose how much time they want to take to do the App. It is recommended that participants make their own routine for using it. The recommended shortest and longest intervention exposure times are: 1 part each day (this will take 19 days to do all of the App), 1 part each week (this will take 19 weeks to do all of the App).
  Interventions: Other: e-health application
- Control Group: Usual Care (No Intervention): Participants in the no intervention Control group continue to get the same care they have been getting (their usual care). The researchers aim to supply the App to participants in both the intervention and control group for a limited time after participation in the study.

INTERVENTIONS:
Other: e-health application — In the first part of this study, an e-health application (MyREADY Transition[TM] BBD App) was developed, targeting the needs of youth with BBD during their transition and transfer from pediatric to adult health care. Program development centered on three core foci of health care transition planning: education, empowerment, and navigation. The intervention has an emphasis on the process of transition in which youth and young adults learn information and develop skills in order to eventually assume maximal responsibility for self-management of their conditions (e.g., learning how to speak directly with health providers) while also providing information to prepare youth for the event of the transfer from pediatric to adult health care.
  Other Names: MyREADY Transition[TM] BBD App
  Arms: Usual Care + MyREADYTransition[TM] BBD App

SUMMARY:
The purpose of this study is to find out if there is a benefit to using the MyREADY Transition[TM] BBD App for brain-based disabilities, compared to not using it. To do this, some of the participants in this study will use the MyREADY Transition[TM] BBD App and others will not use the App. Everyone will continue to get the same care they have been getting (their usual care).

The study team wants to see how youth will use the MyREADY Transition[TM] BBD App as they are getting ready to leave the children's hospital or children's treatment centre. And, they want to see if it will help youth to be knowledgeable about their own health. The study team hopes to see youth taking steps to develop the skills so they become better managers of their health. For example, this would include knowing about their medication or knowing when to ask for help from parents/caregivers and health care providers.

DETAILED DESCRIPTION:
Youth with brain-based disabilities (BBD) see a variety of pediatric doctors and health care providers during their childhood years. Pediatric doctors and care teams are trained to manage the health of children, including physical, behavioural, and mental health issues. Typically by their eighteenth birthday, youth in Canada will need to leave their pediatric doctors and health care providers and go to adult providers instead. Generally, there are more expectations for youth to take charge of their own care when they see an adult care provider. Yet, if youth are not ready for this responsibility, or it is not clear where youth should go for care as adults, their health can sometimes be affected (for example when appointments or medications are missed). We also know that this change can be especially difficult and stressful for youth with BBD and for their families.

In the first part of this project, researchers, healthcare professionals, technology designers, youth and families have worked together to co-create an e-health application called MyREADY Transition[TM] BBD App. In this next part of the project, pediatric health care providers will be asked to share it with their patients who are between 15 and 17 years of age, and who have one of the following conditions: autism spectrum disorder, cerebral palsy, epilepsy, spina bifida, or fetal alcohol spectrum disorder. The MyREADY Transition[TM] BBD App is designed to help youth with health care transition planning, in preparation for their transfer out of the child health system and into the adult health system. The study team wants to see how youth will use the MyREADY Transition[TM] BBD App as they are getting ready to go from pediatric to adult health care services. And, the study team wants to see if it will help them to be more prepared and knowledgeable to manage their own health. The study team hopes to see youth taking steps to be better managers of their health. For example, this would include knowing about their condition or knowing when to ask for help from parents/caregivers and health care providers. After the completion of the study, the researchers will explore the potential to make the App more widely available.

ELIGIBILITY:
Inclusion Criteria:

* Youth with chronological age between 15 and 17 years of age (i.e. before 18th birthday), in one of the four Canadian study regions (Alberta, Ontario, Quebec, Maritimes), followed in pediatric care and for whom a discharge from pediatric care is planned but not for at least 6 months.
* A diagnosis of one of the following neurological brain-based disabilities: autism spectrum disorder, cerebral palsy, epilepsy, spina bifida, or fetal alcohol spectrum disorder.
* Cognitive ability to provide informed consent and the ability to read and understand English or French.
* Access to internet and a smartphone, iPad/tablet or desktop computer.
* TRANSITION-Q score >40 (as a screen to define a minimum threshold for transition readiness based on earlier work).

Exclusion Criteria:

* Youth is in "acute crisis" with unstable physical or mental health that would interfere with the ability to participate in the study.
* Sensory impairments, such as uncorrected vision or hearing loss, which interfere with use of the App intervention.
* Enrolled in a potentially confounding trial (e.g., a different transition intervention study).

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Willem Gorter, MD,PhD,FRCPC, Principal Investigator — McMaster University; Ariane Marelli, MD,MPH,FRCPC, Principal Investigator — McGill University; Adrienne Kovacs, PhD,CPsych, Principal Investigator — Oregon Health and Science University
Locations (9):
- Canada (9):
  - Alberta Health Services and The Governors of the University of Alberta, Edmonton, Alberta
  - Horizon Health Network, Saint John, New Brunswick
  - Izaak Walton Killam Health Centre (IWK), Halifax, Nova Scotia
  - McMaster Children's Hospital, Hamilton Health Sciences, Hamilton, Ontario
  - Lawson Health Research Institute, London, Ontario
  - Children's Hospital of Eastern Ontario Research Institute Inc., Ottawa, Ontario
  - Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Research Institute of the McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gorter JW, Amaria K, Kovacs A, Rozenblum R, Thabane L, Galuppi B, Nguyen L, Strohm S, Mahlberg N, Via-Dufresne Ley A, Marelli A; CHILD-BRIGHT READYorNotTM Brain-Based Disabilities Trial Study Group; CHILD-BRIGHT READYorNot(TM) Brain-Based Disabilities Trial Study Group. CHILD-BRIGHT READYorNot Brain-Based Disabilities Trial: protocol of a randomised controlled trial (RCT) investigating the effectiveness of a patient-facing e-health intervention designed to enhance healthcare transition readiness in youth. BMJ Open. 2021 Mar 26;11(3):e048756. doi: 10.1136/bmjopen-2021-048756. PMID 33771833
- [Derived] Marelli A, Rozenblum R, Bolster-Foucault C, Via-Dufresne Ley A, Maynard N, Amaria K, Galuppi B, Strohm S, Nguyen L, Dawe-McCord C, Putterman C, Kovacs AH, Gorter JW. Development of MyREADY Transition BBD Mobile App, a Health Intervention Technology Platform, to Improve Care Transition for Youth With Brain-Based Disabilities: User-Centered Design Approach. JMIR Pediatr Parent. 2024 Oct 1;7:e51606. doi: 10.2196/51606. PMID 39352737
- See also: Study page on the CHILD-BRIGHT network website — http://www.child-bright.ca/readyornot/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care + MyREADYTransition[TM] BBD App | Control Group: Usual Care
Started | 24 | 28
Completed | 19 | 24
Not Completed | 5 | 4
Not completed — Lost to Follow-up | 4 | 3
Not completed — Only parent outcomes completed | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care + MyREADYTransition[TM] BBD App | Control Group: Usual Care | Total
Number analyzed (Participants) | 24 | 28 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.0 (0.6) | 16.0 (0.8) | 16.0 (0.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Girl/Young woman | 13 | 14 | 27
  Boy/Young man | 9 | 12 | 21
  Other | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: race/ethnicity missing for 2 participants in control group
  Participants
    Ancestry: number analyzed (Participants) | 24 | 26 | 50
    Ancestry: European | 23 | 19 | 42
    Ancestry: East and South Asian | 0 | 2 | 2
    Ancestry: North American Aboriginal | 0 | 2 | 2
    Ancestry: Latin Central and South American | 1 | 0 | 1
    Ancestry: Other | 0 | 3 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Canada: Alberta | 5 | 5 | 10
  Canada: Ontario | 14 | 15 | 29
  Canada: Quebec | 2 | 4 | 6
  Canada: Maritimes | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Transition Readiness Assessment Questionnaire (TRAQ) Change
Description: While Transition Readiness Assessment Questionnaire (TRAQ) measure refinement is ongoing, and other versions are now available, our sample size calculation is based on findings from an intervention trial where the 29-item version of the TRAQ was used. The 29-item version has a Self-management domain score (16 items) and a Self-advocacy domain score (13 items). Both the TRAQ Self-management and TRAQ Self-advocacy domain scores are reported. Scores range from 1 to 5. Higher scores mean better transition readiness.
Time Frame: Baseline and 6-Month Visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care + MyREADYTransition[TM] BBD App | Control Group: Usual Care
Number analyzed (Participants) | 19 | 24
score on a scale
  Self-management Baseline Visit | 2.3 (0.6) | 2.2 (0.5)
  Self-management 6-Month Visit | 2.5 (0.7) | 2.5 (0.9)
  Self-advocacy Baseline visit | 3.4 (0.6) | 3.0 (0.5)
  Self-advocacy 6-Month Visit | 3.6 (0.6) | 3.2 (0.8)

2. Secondary Outcome: Canadian Occupational Performance Measure (COPM) Change
Description: The Canadian Occupational Performance Measure (COPM) is an evidence-based, generic, and individualized outcome measure used to capture a client's self-perception of performance and satisfaction in everyday living over time, by identifying problems in performing activities of daily living. Participants are encouraged to think about things (goals) that they want to do, need to do or are expected to do but can't do, don't do or aren't satisfied with the way they do. Participants are asked to rate current performance using a 10-point scale ranging from 1'not able to do it' to 10 'able to do it very well'. Higher performance scores indicate better perceived performance of the goal. Participants are also asked to rate satisfaction with performance on a 10-point scale ranging from 1 'not satisfied at all' to 10 'extremely satisfied'. Higher satisfaction scores indicate better perceived satisfaction with their performance of the goal.
Time Frame: Baseline and 6-Month Visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care + MyREADYTransition[TM] BBD App | Control Group: Usual Care
Number analyzed (Participants) | 19 | 24
score on a scale
  Performance Baseline Visit | 4.3 (1.8) | 5.3 (2.2)
  Performance 6-Month Visit | 6.0 (1.6) | 6.7 (2.3)
  Satisfaction Baseline Visit | 4.8 (2.1) | 5.2 (2.2)
  Satisfaction 6-Month Visit | 6.3 (1.9) | 7.3 (2.3)

3. Secondary Outcome: TRANSITION-Q Change
Description: The TRANSITION-Q is a 14-item transition readiness/self-management ability scale. This short, clinically meaningful and psychometrically sound scale can be used in research and in pediatric and adolescent clinics to help evaluate readiness for transition to adult care. Item responses ("never" = 0, "sometimes" = 1, and "always" = 2) are summed to create a raw score, with a possible range from 0 to 28. Raw scores are transformed using a table provided by the developers and the transformed scores range from 0-100. A higher score indicates greater transition readiness; exhibiting more self-management skills with higher frequency.
Time Frame: Baseline and 6-Month Visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care + MyREADYTransition[TM] BBD App | Control Group: Usual Care
Number analyzed (Participants) | 19 | 24
score on a scale
  Baseline Visit | 57.0 (10.1) | 56.1 (10.4)
  6-Month Visit | 59.4 (13.2) | 52.2 (19.6)

4. Secondary Outcome: Pediatric Quality of Life Instrument (PedsQL[TM]) Change
Description: The Pediatric Quality of Life Instrument (PedsQL[TM]) takes a modular approach to measuring health-related quality of life (HRQOL) in healthy children and adolescents and those with acute and chronic health conditions. In this study the PedsQL[TM] Pediatric Quality of Life Instrument, Generic Core, Teen Report (13-18 years) was completed. The form is brief (23 items), practical (less than 4 minutes to complete), multidimensional (Physical, Emotional, Social, School Functioning), reliable (Child Self-Report; 0.90) and valid (Distinguishes between healthy children and children with acute and chronic health conditions; distinguishes disease severity within a chronic health condition), and responsive to clinical change over time. Overall Score reported in table, on a 0-100 scale, with higher scores indicating better Health-Related Quality of Life (HRQOL).
Time Frame: Baseline and 6-Month Visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care + MyREADYTransition[TM] BBD App | Control Group: Usual Care
Number analyzed (Participants) | 19 | 24
score on a scale
  Baseline Visit | 64.5 (16.5) | 64.6 (20.8)
  6 Month Visit | 63.2 (18.3) | 66.2 (18.1)

5. Secondary Outcome: Measure of Process of Care (MPOC) Change
Description: The Measure of Processes of Care (MPOC) is a well-validated and reliable self-report measure of parents' perceptions of the extent to which the health services they and their children receive are family-centred. The original version of MPOC is a 56-item questionnaire; as of 1999 there is a shorter, 20-item version called MPOC-20 which was used (and modified with permission) in this study. Five MPOC-20 scale scores are reported: Enabling and Partnership, Providing General Information, Providing Specific Information, Coordination and Comprehensive Care, Respectful and Supportive Care. A 7-point scale is used, ranging from 7 "to a very great extent", 6 = "to a great extent", 5 = "to a fairly great extent", 4 = "to a moderate extent", 3 = "to a small extent", 2 = "to a very small extent", and 1 = "not at all". A score of 0 indicates "not applicable". Higher MPOC-20 scale scores indicate better family-centred care.
Time Frame: Baseline and 6-Month Visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care + MyREADYTransition[TM] BBD App | Control Group: Usual Care
Number analyzed (Participants) | 19 | 24
score on a scale
  Enabling and Partnership Baseline Visit | 4.6 (1.5) | 4.3 (1.6)
  Enabling and Partnership 6-Month Visit | 4.5 (1.8) | 4.4 (1.7)
  Providing General information Baseline Visit | 3.4 (1.6) | 3.6 (1.7)
  Providing General information 6 Month Visit | 3.3 (1.7) | 3.6 (1.8)
  Providing Specific information Baseline Visit | 4.2 (1.5) | 4.3 (1.4)
  Providing Specific information 6-Month Visit | 4.2 (2.1) | 4.4 (1.6)
  Coordination and comprehensive care Baseline Visit | 4.8 (1.5) | 4.7 (1.3)
  Coordination and comprehensive care 6-Month Visit | 4.6 (2.0) | 4.7 (1.6)
  Respectful and supportive care Baseline Visit | 5.1 (1.1) | 5.1 (1.1)
  Respectful and supportive care 6-Month Visit | 4.8 (1.6) | 4.9 (1.5)

6. Secondary Outcome: Health Utilities Index® (Hui2/3) Proxy-Assessed Change
Description: The HUI is a generic health status instrument developed in Canada for use with children and has been incorporated in numerous clinical studies as well as the Canadian Community Health Survey, allowing the generation of norms for most age groups. The HUI Mark II includes 7 attributes: Sensation, Mobility, Emotion, Cognition, Self-care, Pain and Fertility with each attribute divided into 3 to 5 levels. The HUI III includes 8 attributes: Vision, Hearing, Speech, Ambulation, Dexterity, Emotion, Cognition and Pain. Each attribute of the HUI III consists of 5 to 6 levels. We report the overall health rating at Baseline and 6-Month Visit measured on a scale from 1 (Poor) to 5 (Excellent)
Time Frame: Baseline and 6-Month Visit
Population: 1. overall health rating missing at both Baseline and 6-Month Visit in Control Group: Usual Care Arm.
  2. overall health ratings missing at 6-Month visit in Usual Care + MyREADYTransition[TM] BBD App Arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care + MyREADYTransition[TM] BBD App | Control Group: Usual Care
Number analyzed (Participants) | 19 | 24
units on a scale
  Baseline Visit: number analyzed (Participants) | 19 | 23
  Baseline Visit | 3.9 (0.9) | 4.1 (1.0)
  6-Month Visit: number analyzed (Participants) | 17 | 23
  6-Month Visit | 4.0 (0.8) | 4.0 (0.7)

7. Secondary Outcome: Resource Use Questionnaire (RUQ) Change
Description: The RUQ is typically an interviewer-administered questionnaire for parents of children aged 11 to 18 years. The original RUQ measures the family resource use of condition-related treatments, services and programs, as well as parent time losses and family out-of-pocket costs. It also documents condition-related government subsidies and funding that families receive. Resources measured include those delivered by a parent, by other providers (e.g. behavioural specialist) or a combination of both. In this project, we will use a modified subset of RUQ questions, self-completed by the parent/caregiver. We report information collected at the 6-Month Visit about the number of participants in each arm who reported any hospitalizations during the study.
Time Frame: 6-Month Visit
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care + MyREADYTransition[TM] BBD App | Control Group: Usual Care
Number analyzed (Participants) | 19 | 24
Participants | 2 | 3

8. Secondary Outcome: System Usability Scale (SUS)
Description: The SUS will be administered to youth in the Experimental Arm. The measure focus is on users' utilization of the application and its features, the perceived value and their experience and satisfaction with the intervention. The self-reported survey will provide additional information about the users' adherence, behavior, motivation and experience with the IT platform, as well as about the main reasons for using or not using it. Measures youth's subjective perceptions of the usability of the App, scored from 0 - 100 with a higher score indicating greater usability.
Time Frame: 6-Month Visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care + MyREADYTransition[TM] BBD App
Number analyzed (Participants) | 18
score on a scale | 65.4 (26.8)

9. Other Pre Specified Outcome: Utilization of Intervention (Usage, Adherence, and Fidelity)
Description: Mixed methods will be used to assess MyREADY Transition[TM] BBD App usage, adherence and fidelity, and to identify the barriers and facilitators to using the e-health application for users. Quantitative data will be collected through participant self-report and by the app daily through study completion. For a subset of participants in the intervention group, qualitative data will be collected via interview. Utilization of Intervention reporting at 6-Month Visit.
  Usage reported here as the average number of times intervention participants logged into the App.
Time Frame: 6-Month Visit
Population: Average number of times intervention group participants logged into the App intervention. Indicates App intervention access or engagement. Higher scores indicate better engagement.
Measure: Mean (Standard Deviation); unit: times
Arm/Group | Usual Care + MyREADYTransition[TM] BBD App
Number analyzed (Participants) | 24
times | 11.2 (9.5)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Usual Care + MyREADYTransition[TM] BBD App | Control Group: Usual Care
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/24
Other Adverse Events (participants affected / at risk) | 0/19 | 0/24

LIMITATIONS AND CAVEATS:
The planned sample size was 264; 43 participants completed follow-up. With significant start-up delays and recruitment curtailed by the COVID-19 pandemic, the limited feasibility to recruit our sample ultimately led to the early stop of the trial. As approved by ethics, we dropped the health economic outcome analysis (Health card number linking, Health Utilities Index (HUI), Resource Use Questionnaire (RUQ)) and destroy stored health card number data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-09): https://cdn.clinicaltrials.gov/large-docs/50/NCT03852550/Prot_SAP_000.pdf